CLINICAL TRIAL: NCT00679783
Title: Phase II, Open Label, Non-Randomized Study of AZD2281 in the Treatment of Patients With Known BRCA or Recurrent High Grade Serous/ Undifferentiated Tubo-Ovarian Carcinoma and in Known BRCA or Triple Negative Breast Cancer to Determine Response Rate and Correlative Markers of Response
Brief Title: Phase II Study of AZD2281 in Patients With Known BRCA Mutation Status or Recurrent High Grade Ovarian Cancer or Patients With Known BRCA Mutation Status/ Triple Neg Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00020
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Carcinoma; Breast Cancer
Keywords: Breast cancer; Ovarian cancer; BRCA; Triple negative; Poly(ADP ribose) polymerases; Known BRCA or Recurrent High Grade Serious/ Undifferentiated Tubo- Ovarian Carcinoma; Known BRCA or Triple Negative Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: 4 parallel arms for the 2 tumour types and the BRCA mutation groups:
  1. Triple negative breast Cancer with unknown BRCA mutation status: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally
  2. Known BRCA mutation positive breast cancer: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) to be administered orally
  3. High grade serous/undifferentiated tubo-ovarian carcinoma with unknown BRCA status: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally
  4. Known BRCA mutation positive ovarian cancer: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally.
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Triple negative breast Cancer with unknown BRCA mutation status: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally
  AZD2281, PARP inhibitor Olaparib tablets, oral
  Interventions: Drug: AZD2281
- 2 (Experimental): Known BRCA mutation positive breast cancer: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) to be administered orally
  AZD2281, PARP inhibitor Olaparib tablets, oral
  Interventions: Drug: AZD2281
- 3 (Experimental): High grade serous/undifferentiated tubo-ovarian carcinoma with unknown BRCA status: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally
  AZD2281, PARP inhibitor Olaparib tablets, oral
  Interventions: Drug: AZD2281
- 4 (Experimental): Known BRCA mutation positive ovarian cancer: AZD2281 400 mg bid (capsules)/ 300 mg bid (tablets) administered orally
  AZD2281, PARP inhibitor Olaparib tablets, oral
  Interventions: Drug: AZD2281

INTERVENTIONS:
Drug: AZD2281 — PARP inhibitor Olaparib tablets, oral
  Other Names: Olaparib

SUMMARY:
This is a Phase II, open label, non randomized correlative study of AZD2281 in patients with recurrent breast and ovarian cancer in both BRCA inherited mutation carriers and non-carriers to identify objective response rate and to assess for early markers of activity and to assess correlative markers that may provide helpful information for subsequent clinical trials. Approximately 110 patients from 7 centers in Canada will be enrolled into this study

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade serous and/or undifferentiated carcinoma of ovary, fallopian tube or peritoneum
* Oestrogen, progesterone and HER2 negative advanced adenocarcinoma of the breast
* Known BRCA positive breast cancer or ovarian cancer, that is not high grade serous or undifferentiated tubo-ovarian carcinoma.
* Performance status of no more than 2.

Exclusion Criteria:

* Any chemotherapy, radiotherapy ( except palliative), endocrine or immunotherapy within 4 weeks prior to entry
* Major surgery with 4 weeks of entering the study and must have recovered from effects of any major surgery .

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-07-08 (Actual); Primary Completion 2010-03-26 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gelmon, MD, Study Chair — British Columbia Cancer Agency; Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca
Locations (6):
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Ang JE, Gourley C, Powell CB, High H, Shapira-Frommer R, Castonguay V, De Greve J, Atkinson T, Yap TA, Sandhu S, Banerjee S, Chen LM, Friedlander ML, Kaufman B, Oza AM, Matulonis U, Barber LJ, Kozarewa I, Fenwick K, Assiotis I, Campbell J, Chen L, de Bono JS, Gore ME, Lord CJ, Ashworth A, Kaye SB. Efficacy of chemotherapy in BRCA1/2 mutation carrier ovarian cancer in the setting of PARP inhibitor resistance: a multi-institutional study. Clin Cancer Res. 2013 Oct 1;19(19):5485-93. doi: 10.1158/1078-0432.CCR-13-1262. Epub 2013 Aug 6. PMID 23922302
- [Derived] Gelmon KA, Tischkowitz M, Mackay H, Swenerton K, Robidoux A, Tonkin K, Hirte H, Huntsman D, Clemons M, Gilks B, Yerushalmi R, Macpherson E, Carmichael J, Oza A. Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triple-negative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol. 2011 Sep;12(9):852-61. doi: 10.1016/S1470-2045(11)70214-5. Epub 2011 Aug 19. PMID 21862407
- See also: D0810C00020_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=194&filename=D0810C00020.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on July 8, 2008 and efficacy and safety data were collected up to the data cut-off of March 26, 2010. Patients were enrolled at 6 centres in Canada. Of the 112 patients who gave informed consent 21 patients failed eligibility criteria or withdrew their consent and were not allocated to treatment.
Pre-assignment Details: The study enrolled both known BRCA mutation carriers and patients with unknown BRCA status. Those with unknown status at entry had to provide a DNA sample for BRCA. One participant in arm 4 discontinued before receiving study drug and is excluded from the safety analysis set mutation analysis. Study data are summarised by confirmed mutation status.
Groups:
- BRCA Positive Non-serous Ovarian: Patients with non-serous ovarian cancer who have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2. (Serous tumors are the most common subtype of ovarian cancer; other subtypes are grouped together as "non-serous" in this study).
- BRCA Positive Serous Ovarian: Patients with serous ovarian cancer who have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2. (Serous tumors are the most common subtype of ovarian cancer).
- BRCA Negative Non-serous Ovarian: Patients with non-serous ovarian cancer who do not have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2
- BRCA Negative Serous Ovarian: Patients with serous ovarian cancer who do not have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2
- BRCA Positive Non-triple Negative Breast: Patients with non-Triple negative breast cancer (non-TNBC) who have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2. Non-TNBC are cancers that have receptors for oestrogen, progesterone or Her2
- BRCA Positive Triple Negative Breast: Patients with Triple negative breast cancer (TNBC) who have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2. TNBC are cancers that don't have receptors for oestrogen, progesterone or Her2 (Some commonly used breast cancer treatments don't work for TNBC)
- BRCA Negative Triple Negative Breast: Patients with Triple negative breast cancer (TNBC) who do not have a harmful mutation in the "breast cancer genes" BRCA1 or BRCA2.
Period: Overall Study
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Started | 4 (Gave Informed consent and passed screening) | 13 (Gave Informed consent and passed screening) | 3 (Gave Informed consent and passed screening) | 45 (Gave Informed consent and passed screening) | 5 (Gave Informed consent and passed screening) | 5 (Gave Informed consent and passed screening) | 16 (Gave Informed consent and passed screening)
Completed | 2 (Patients who discontinued treatment following disease progression.) | 10 (Patients who discontinued treatment following disease progression.) | 2 (Patients who discontinued treatment following disease progression.) | 25 (Patients who discontinued treatment following disease progression.) | 4 (Patients who discontinued treatment following disease progression.) | 5 (Patients who discontinued treatment following disease progression.) | 15 (Patients who discontinued treatment following disease progression.)
Not Completed | 2 | 3 | 1 | 20 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Not Captured | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Ongoing at data cut-off | 2 | 2 | 0 | 9 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast | Total
Number analyzed (Participants) | 4 | 13 | 3 | 44 | 5 | 5 | 16 | 90
Age, Continuous [Mean (Standard Deviation); unit: Year] | 60 (18.7) | 53.7 (7.3) | 60.3 (12.9) | 61 (9.5) | 49.4 (20.5) | 44.8 (15.5) | 48.8 (5.5) | 52.9 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 3 | 44 | 5 | 5 | 16 | 90
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Evaluated According to Response Evaluation Criteria In Solid Tumors (RECIST) Guidelines
Description: Percentage of participants with confirmed best RECIST response of complete response (CR) or partial response (PR). Patients with a best RECIST response of CR or PR had to have a confirmed response at least 28 days later.
Time Frame: Each patient with measurable disease at baseline was assessed for Objective Response from the sequence of RECIST scan data up to data cut-off, 26 March 2010. RECIST scans were performed every 8 weeks (+/- 2 weeks) from randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 4 | 13 | 3 | 43 | 4 | 4 | 15
Percentage of participants | 75 [30.06 to 95.44] | 30.77 [12.68 to 57.63] | 0 [0 to 56.15] | 25.58 [14.93 to 40.24] | 0 [0 to 48.99] | 0 [0 to 48.99] | 0 [0 to 20.39]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with confirmed best Response Evaluation Criteria In Solid Tumours (RECIST) response of complete response (CR), partial response (PR) orStable Disease (SD)
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 4 | 13 | 3 | 44 | 5 | 5 | 16
Percentage of participants | 75 [30.06 to 95.44] | 53.85 [29.14 to 76.79] | 0 [0 to 56.15] | 47.73 [33.75 to 62.06] | 60 [23.07 to 88.24] | 20 [3.62 to 62.45] | 0 [0 to 19.36]

3. Secondary Outcome: Duration of Response
Description: Duration of response is measured from the time the measurement criteria for CR or PR are met (whichever is first recorded) until the patient progresses (per RECIST criteria). If patient did not progress, they are censored at their last objective tumour assessment date.
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomization (+/- 2 weeks) until data cut-off on 26 March 2010.
Measure: Median (Full Range); unit: Days
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 3 | 4 | 0 | 11 | 0 | 0 | 0
Days | 277 [261 to 504] | 113 [109 to 446] |  | 384 [105 to 396] |  |  |

4. Secondary Outcome: Best Percentage Change From Baseline in Tumour Size
Description: The best percentage change (reduction) from baseline in tumour size (defined as the sum of the longest diameters as measured among all target lesions).
Time Frame: Each patient with measurable disease at baseline was assessed for best percentage change in tumour size from the sequence of RECIST scan data up to data cut-off, 26 March 2010. RECIST scans were performed every 8 weeks (+/- 2 weeks) from randomization.
Measure: Median (Full Range); unit: Percentage
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 4 | 13 | 2 | 38 | 4 | 4 | 14
Percentage | -44.5 [-64 to 4] | -21.6 [-100 to 16] | 33.6 [14 to 53] | -14.1 [-95 to 83] | -35.3 [-48 to 10] | -36.4 [-50 to 11] | 21.3 [-3 to 50]

5. Secondary Outcome: CA-125 Levels (Ovarian Cancer Patients Only)
Description: A response according to CA-125 has occurred if there is at least a 50% reduction in CA-125 levels from a pre-treatment sample.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 4 | 12 | 3 | 35 | 0 | 0 | 0
Percentage of participants | 75 [30.06 to 95.44] | 33.33 [13.81 to 60.94] | 0 [0 to 56.15] | 28.57 [16.33 to 45.05] |  |  |

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose to the earlier date of radiologic progression (as per Response Evaluation Criteria In Solid Tumours (RECIST) criteria or death by any cause in the absence of objective progression.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Number analyzed (Participants) | 4 | 13 | 3 | 44 | 5 | 5 | 16
Days | 346.5 [51 to 553] | 219 [1 to 503] | 79.5 [1 to 109] | 192 [1 to 559] | 165 [53 to 168] | 106 [37 to 277] | 54 [1 to 111]

ADVERSE EVENTS:
Description: One participant in arm 4 discontinued before receiving study drug and is excluded from the safety analysis set mutation analysis
Arm/Group | BRCA Positive Non-serous Ovarian | BRCA Positive Serous Ovarian | BRCA Negative Non-serous Ovarian | BRCA Negative Serous Ovarian | BRCA Positive Non-triple Negative Breast | BRCA Positive Triple Negative Breast | BRCA Negative Triple Negative Breast
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/13 | 0/3 | 6/44 | 0/5 | 2/5 | 2/16
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13 | 3/3 | 44/44 | 5/5 | 5/5 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRCA Positive Non-serous Ovarian (N=4) | BRCA Positive Serous Ovarian (N=13) | BRCA Negative Non-serous Ovarian (N=3) | BRCA Negative Serous Ovarian (N=44) | BRCA Positive Non-triple Negative Breast (N=5) | BRCA Positive Triple Negative Breast (N=5) | BRCA Negative Triple Negative Breast (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin Decreased (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hernia Repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BRCA Positive Non-serous Ovarian (N=4) | BRCA Positive Serous Ovarian (N=13) | BRCA Negative Non-serous Ovarian (N=3) | BRCA Negative Serous Ovarian (N=44) | BRCA Positive Non-triple Negative Breast (N=5) | BRCA Positive Triple Negative Breast (N=5) | BRCA Negative Triple Negative Breast (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 9 | 2 | 28 | 3 | 5 | 8
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1 | 18 | 2 | 3 | 4
Abdominal Distension (Gastrointestinal disorders) | 2 | 3 | 0 | 11 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 11 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 11 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 0 | 5 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 5 | 0 | 5 | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 0 | 5 | 0 | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 12 | 1 | 28 | 3 | 3 | 7
Oedema Peripheral (General disorders) | 2 | 3 | 0 | 8 | 0 | 0 | 2
Chills (General disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Axillary Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1
Secretion Discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 7 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Breast Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vulvovaginitis Streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Tooth Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight Decreased (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 4 | 0 | 0 | 0
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Glucose Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Iron Decreased (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Murmur (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram Qt Prolonged (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 7 | 1 | 13 | 2 | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 6 | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 4 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2 | 1 | 1 | 3
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 1 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 5 | 1 | 9 | 2 | 2 | 0
Headache (Nervous system disorders) | 3 | 2 | 0 | 7 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 6 | 1 | 5 | 1 | 1 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental Impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 7 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Genital Rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic Discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 5 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 5 | 2 | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 6 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less